CLINICAL TRIAL: NCT00707577
Title: A Randomized Controlled Trial of a Maintenance Program for the Be Fit Employee Wellness Program at Massachusetts General Hospital
Brief Title: A Maintenance Program for the Be Fit Employee Wellness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007p001384; K23HL093221 (NIH)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Overweight
Keywords: Worksite Wellness; Weight loss and maintenance; Physical Activity; Health and Fitness interventions; Healthy eating; Weight loss; Maintenance programs
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based maintenance program (Experimental): 9-month Internet based self-monitoring maintenance program to track weight, exercise, and food logs
  Interventions: Behavioral: Internet-based maintenance program
- Control (No Intervention): No maintenance program provided

INTERVENTIONS:
Behavioral: Internet-based maintenance program — The Be Fit maintenance program is a randomized controlled trial of a 9 month intervention to maintain weight loss and physical activity after completion of the 12 week wellness program. Six teams of 25 participants will be randomized to the intervention or to usual care. There are 2 key elements to the maintenance program: personal contact and Internet contact. The personal contact enables the participants to continue receiving face-to-face support from a Be Fit nutritionist and trainer. The Internet interface is an opportunity for the participants to self-monitor their own progress while still under the guidance of the program.
  Arms: Internet-based maintenance program

SUMMARY:
This research study is being done: 1) to determine if the MGH Be Fit program helps employees to change their nutrition and exercise habits and lower their risk for chronic diseases, such as heart disease and diabetes and 2) to determine if a maintenance program following the Be Fit 12 week program will help employees to keep the positive health changes.

DETAILED DESCRIPTION:
The main objectives of this trial are to determine if employees who participate in the Be Fit 12 week program and are randomized to a 9 month maintenance program are more likely to maintain weight loss, physical activity level, and reduction of other clinical risk factors for disease compared to the control group. Secondary objectives are to determine if employees who participate in the maintenance intervention have fewer chronic diseases related to lifestyle factors and lower health care costs at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* MGH (benefited) employees who enroll in the Be Fit program
* Able to commit to 1 year of active research participation

Exclusion Criteria:

* Not enrolled in the Be Fit program
* Decline participation in the research study
* Withdrawal from the Be Fit 12 week program prior to completion
* Women who are currently pregnant or suspect they may be pregnant
* Plans to leave MGH within 3 months from enrolling in Be Fit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2008-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Thorndike AN, Sonnenberg L, Healey E, Myint-U K, Kvedar JC, Regan S. Prevention of weight gain following a worksite nutrition and exercise program: a randomized controlled trial. Am J Prev Med. 2012 Jul;43(1):27-33. doi: 10.1016/j.amepre.2012.02.029. PMID 22704742

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Internet-based Maintenance Program | Control
Started | 174 | 156
Completed | 120 | 118
Not Completed | 54 | 38
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 34 | 25
Not completed — Left employment | 13 | 10
Not completed — Pregnancy | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet-based Maintenance Program | Control | Total
Number analyzed (Participants) | 174 | 156 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.8) | 41.6 (13.6) | 42.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 123 | 280
  Male | 17 | 33 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  White | 148 | 124 | 272
  Non-white | 26 | 32 | 58
Region of Enrollment [Number; unit: participants]
  United States | 174 | 156 | 330
Married or living with significant other [Count of Participants; unit: Participants] | 110 | 83 | 193
Employment at MGH > 5 years [Count of Participants; unit: Participants] | 89 | 69 | 158
BMI greater than 25 [Count of Participants; unit: Participants] | 115 | 95 | 210
Current smoking [Count of Participants; unit: Participants] | 9 | 6 | 15
Amount of physical activity/week [Median (Inter-Quartile Range); unit: hours] | 2.6 [1 to 6.0] | 3.5 [1 to 5.8] | 3.0 [1 to 6.0]

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Mean number of pounds lost at the end of the 10-week program and 9-month maintenance program
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Internet-based Maintenance Program | Control
Number analyzed (Participants) | 157 | 145
pounds | 3.4 (8.8) | 2.5 (8.8)
Statistical Analysis 1: Comparison: Internet-based Maintenance Program vs Control; Test type: Superiority; p < 0.05, Regression, Linear; random effects regression models for panel data adjusted for clustering within team

ADVERSE EVENTS:
Arm/Group | Internet-based Maintenance Program | Control
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/156
Other Adverse Events (participants affected / at risk) | 0/174 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No